CLINICAL TRIAL: NCT07301658
Title: Evaluation of the Effectiveness and Safety of Revodiol Calming Cream® in the Management of Atopic Dermatitis Under Dermatological Control.
Brief Title: Efficacy and Safety of Revodiol Calming Cream® in Atopic Dermatitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Centro Médico Complutense Grupo Virtus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: caCBD
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dermatitis efficacy test under dermatological control (Experimental)
  Interventions: Other: Novel dermocosmetic product containing cannabidiol (CBD) and Annona cherimola fruit extract.
- Dermatitis efficacy test under dermatological control and pediatric supervision (Experimental)
  Interventions: Other: Novel dermocosmetic product containing cannabidiol (CBD) and Annona cherimola fruit extract.

INTERVENTIONS:
Other: Novel dermocosmetic product containing cannabidiol (CBD) and Annona cherimola fruit extract. — Apply twice a day on the affected skin area to protect it, previously cleaned and dried. No rinsing is required. Volunteers were instructed not to use any other cosmetic product in the study area until the end of the study.

SUMMARY:
A 56-day clinical study evaluated Revodiol Calming Cream on pediatric and adult participants with mild to moderate atopic-prone skin under dermatological supervision. The product was applied twice daily, and efficacy was assessed through dermatological scoring, instrumental measurements, and subjective questionnaires. Results aimed to show improvements in barrier function, hydration, skin texture, and reduction of erythema, dryness, and pruritus, with feedback on comfort and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Sex: both.
* Age: from 0 months onwards (includes children and adults).
* Atopic-prone skin.
* Mild to moderate flare-up.
* Skin dryness.
* Signed informed consent (by the volunteer or legal guardian as applicable).
* Adequate understanding of the clinical study by the participant or legal guardian.
* Good physical and psychological health.
* No application of any product on the experimental area on the first day of the trial.
* Availability to guarantee visits to the research center.

Exclusion Criteria:

* History of allergies to cosmetic products.
* Recent surgery or treatments in the study area.
* Oncology patients.
* Use of antihistamines and antibiotics within 15 days prior to the start of the study.
* Treatment with antihistamines, antibiotics, corticosteroids, immunosuppressants or completion of such treatment within 15 days prior to the start of the study.
* Use of any other product for dermatitis during the study.
* Sun exposure or UVA rays during the study.
* Participation in another clinical study.
* Health problems that may compromise adherence to the study protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
SCORAD (SCORing Atopic Dermatitis) Index | 56 days
  The assessment with the SCORAD index included lesion extent and the intensity of objective parameters such as erythema, edema/papules, exudation/crusting, lichenification, excoriation, and dryness, as well as subjective symptoms including pruritus and sleep disturbance. The scale evaluates symptoms from 0 (no signs) to 3 (severe).

SECONDARY OUTCOMES:
Biometric Analysis | 56 days
  Using Mexameter® MX 18 probe anti-erythema efficacy was determined by measuring the light reflected by the skin .
Biometric Analysis | 56 days
  Cutaneous topography was evaluated using the Visioscan®
Biometric Analysis | 56 days
  Skin barrier function efficacy was determined by measuring the transepidermal water loss (TEWL) using the Tewameter® TM 300 probe .
Biometric Analysis | 56 days
  Skin renewal efficacy was determined by measuring skin desquamation using Corneofix® F 20 sheets.
Subjective evaluation | 56 days
  In adult participants, quality of life was assessed using the validated Dermatology Life Quality Index (DLQI) questionnaire. The DLQI consists of 10 items covering symptoms, daily activities, leisure, work/school, personal relationships, and treatment.
Adverse events record | 28 and 56 days
  Adverse events record
Tolerance evaluation | 56 days
  At the end of the study, the dermatologist assessed local tolerance based on the presence and intensity (mild, moderate, severe) of erythema, xerosis/desquamation, oedema, exudation, comedogenicity, and pigmentation alterations. Causality was also rated according to the scale: not related, improbable, possible, probable, certain, or not assessable.

CONTACTS AND LOCATIONS:
Locations (1):
- i+Med S.Coop., Vitoria-Gasteiz, Álava, Spain

IPD SHARING:
Plan to Share IPD: No